CLINICAL TRIAL: NCT01756222
Title: Bicuspid Aortic Valve and Ascending Aortic Aneurysm Registry
Brief Title: Bicuspid Aortic Valve (BAV) Registry
Acronym: BAV
Status: Recruiting | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Dr. Bo Yang, MD, University of Michigan
Other Study IDs: HUM00035836
Record Dates: First submitted 2012-12-19; First posted 2012-12-25 (Estimated); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Bicuspid Aortic Valve
Keywords: Bicuspid Aortic Valve Disease; Bicuspid Aortic Valve; BAV
MeSH Terms: conditions — Bicuspid Aortic Valve Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (1):
- Bicuspid Aortic Valve Disease Patients: Patients with the diagnosis of BAV disease.

SUMMARY:
The purpose of this registry is to gather information on patients with bicuspid aortic valve disease.

DETAILED DESCRIPTION:
The purpose of this registry is to gather information on patients with bicuspid aortic valve disease. The data collected in the registry will be used to assess patterns of aortic dilation, responses to medical therapy based on serial imaging and to assess for potential genetic markers of this disease

ELIGIBILITY:
Inclusion Criteria:

* Any patient over the age of 18 who is able/willing to give informed consent with the diagnosis of bicuspid aortic valve disease, a family history of this disease or an ascending aortic aneurysm that is idiopathic can be included in the registry.

Exclusion Criteria:

* Patients unable or unwilling to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary clinic
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2010-04; Primary Completion 2040-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Characterizing patients with bicuspid aortic valve disease | 30 years
  Identifying patients with bicuspid aortic valve disease, assessing the effect of medical intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Yang, MD, Principal Investigator — University of Michigan
Locations (1):
- Univeristy of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided